CLINICAL TRIAL: NCT02427074
Title: Comparative Study Between Radiofrequency and Balloon Compression of the Gasserian Ganglion in the Treatment of Idiopathic Trigeminal Neuralgia
Brief Title: Comparison Between Radiofrequency and Balloon Compression in the Treatment of Idiopathic Trigeminal Neuralgia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted due to futility
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Hugo Sterman Neto, medical doctor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1180/09
Record Dates: First submitted 2015-04-18; First posted 2015-04-27 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balloon Compression Rhizotomy (Active Comparator): Patients that are submitted to Balloon Compression Rhizotomy
  Interventions: Procedure: Balloon Compression Rhizotomy
- Radiofrequency Thermal Coagulation Rhizotomy (Active Comparator): Patients that are submitted to Radiofrequency Thermal Coagulation Rhizotomy
  Interventions: Procedure: Radiofrequency Thermal Coagulation Rhizotomy

INTERVENTIONS:
Procedure: Balloon Compression Rhizotomy — The balloon compression rhizotomy is performed in a percutaneous fashion where a Fogarty catheter is positioned in the gasserian ganglion and inflated with 0,7 milliliters of radiopaque dye during 120 seconds.
  Arms: Balloon Compression Rhizotomy
Procedure: Radiofrequency Thermal Coagulation Rhizotomy — The gasserian ganglion is submitted to a controlled thermal coagulation with a electrode with 80 Celsius degrees of temperature during 60 seconds on the specific division.
  Arms: Radiofrequency Thermal Coagulation Rhizotomy

SUMMARY:
Two percutaneous procedures used in the treatment of idiopathic trigeminal neuralgia are analysed. The effects on pain relief, alterations in cutaneous sensibility and olfactory and salivatory functions are analysed as well.

DETAILED DESCRIPTION:
Patients diagnosed with idiopathic trigeminal neuralgia, refractory or intolerant to medical treatment, are randomly assigned (after signing a consent form), to receive one of two percutaneous procedures. The patients are evaluated a week before and a week, a month, two months, three months and six months after the surgery.

The questionnaires (Short-Form of the McGill Pain Questionnaire - SF-MPQ, Douleur Neuropathique - DN4, Neuropathic Pain Symptom Inventory - NPSI, Brief Pain Inventory - BPI, Global Clinical Impression - GCI, Hospital Anxiety and Depression - HAD, Brief World Health Organization Quality of Life Questionnaire - WHOQOL-brief, Pain Catastrophizing Scale - PCS) and tests (Quantitative Sensory Testing - QST, olfactory threshold - OT - and discrimination - OD, taste threshold - TT, and salivatory quantification - SQ) are applied as follows:

* Pre-op evaluation: SF-MPQ, DN4, BPI, NPSI, HAD, WHOQOL-brief, PCS, QST, OT, OD, TT, SQ.
* First visit post-op: SF-MPQ, BPI, NPSI, GCI
* Second visit post-op: SF-MPQ, BPI, NPSI, GCI
* Third visit post-op: SF-MPQ, BPI, NPSI, GCI
* Fourth visit post-op: SF-MPQ, DN4, BPI, NPSI, GCI, WHOQOL-brief, HAD, PCS, QST, OT, TT, SQ.
* Fifth visit post-op: SF-MPQ, DN4, BPI, NPSI, GCI, WHOQOL-brief, HAD, PCS, QST, OT, OD, TT, SQ.

Patients with pain recurrence are excluded after the last visit attended. An exploratory analysis is made with 30 patients for a proper sample size calculation during the study.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Trigeminal Neuralgia
* Refractory/Intolerable medical treatment
* Pain restricted to second or third trigeminal division

Exclusion Criteria:

* Secondary Trigeminal Neuralgia
* Pain restricted to the first trigeminal division
* Refuse to participate
* Unable to comprehend the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Pain relief using numeric rating scale | 6 months
  Worst pain in the last 24h scale in the Brief Pain Inventory

SECONDARY OUTCOMES:
Changes in how the pain is perceived by the patient assessed by the Short-Form of the McGill Pain Questionnaire | 6 months
  Short-Form of the McGill Pain Questionnaire
Changes in neuropathic pain quality assessed by Douleur Neuropatique 4 | 6 months
  Douleur Neuropatique 4
Evaluation of chronic pain and its influence in patients life assessed by Brief Pain Inventory | 6 months
  Brief Pain Inventory
Changes in types of symptoms of neuropathic pain assessed by Neuropathic Pain Symptom Inventory | 6 months
  Neuropathic Pain Symptom Inventory
Changes in quality of life assessed by World Health Organization Quality of Life - brief form | 6 months
  World Health Organization Quality of Life - brief form
Both patient and investigator impression in the treatment assessed by Global Clinical Impression | 6 months
  Global Clinical Impression
Evaluation of how pain affects patients perception assessed by Pain Catastrophizing Scale | 6 months
  Pain Catastrophizing Scale
Onset of changes in anxiety or depression assessed by Hospital Anxiety and Depression | 6 months
  Hospital Anxiety and Depression
Quantification of facial sensibility changes assessed by Quantitative Sensorial Testing | 6 months
  Quantitative Sensorial Testing
Changes in olfactory threshold assessed by isopropanol solution | 6 months
  Olfactory Threshold using isopropanol solution
Changes in gustatory threshold assessed using sweet, sour, salty and bitter solutions | 6 months
  Gustatory Threshold using sweet, sour, salty and bitter solutions
Changes in salivary flow assessed using cotton weights | 6 months
  Evaluation of salivary flow using cotton weights
Changes in olfactory discrimination assessed using Sniffin' Sticks | 6 months
  Using Sniffin' Sticks to evaluate olfactory discrimination

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ciampi, MD, PhD, Study Chair — HCFMSUP
Locations (1):
- HCFMSUP, São Paulo, São Paulo, Brazil